CLINICAL TRIAL: NCT04562246
Title: Laboratory Validation of SARS-CoV-2 IgG and IgM Serologic Assays on an Automated Immunoassay System
Brief Title: SARS-CoV-2 IgG and IgM Serologic Assays
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Bernard Cook, Division Head, Chemistry-Pathology, Henry Ford Health System
Other Study IDs: 13839
Record Dates: First submitted 2020-09-22; First posted 2020-09-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PCR positive subjects: Patients who receive positive test result from RT-PCR for SARS-CoV-2.
  Interventions: Diagnostic Test: Serologic assays for antibodies to SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: Serologic assays for antibodies to SARS-CoV-2 — Beckman Coulter and Roche automated immunoassays

SUMMARY:
The primary objective is to assess and validate the ability of the Beckman Coulter Access COVID-19 IgG and IgM assays to detect immunity in COVID-19 patients in the Henry Ford Hospital Health System.

DETAILED DESCRIPTION:
Overview: The design validation strategy for this study is to validate the detection of COVID-19 antibodies in subjects at Henry Ford Health System (HFHS) who test negative or positive with RT-PCR for SARS-CoV-2 using a fully automated system. This is a study of the immune response of subjects who have recovered from COVID-19 infection.

Methods: There are now commercial testing products from major invitro diagnostic diagnostics companies that appear to have been developed with significantly greater test performance in mind. HFHS (HFHS) intends to make this testing available in the near future after a rigorous verification of analytical performance. This verification will be done in collaboration a with select and proven IVD partner.

All HFHS patients > 18 years of age who were evaluated and who have COVID-19 PCR test results will have their medical records studies and a left-over specimen tested for validation purposes. This validation study will begin May 15, 2020 through November 15, 2020.

Impact: IVD manufacturers must rely on test specimens from suppliers (typically hospitals and reference laboratories) and attempt to replicate the test performance that will be achieved in the actual medical testing environment. In fact, samples collected and provided to vendors are usually at the convenience of the supplying institution. Data on the real-world performance of COVID-19 antibody tests derived from this study will have significant implications for patients and health systems, including patient disposition, risk prediction, return to work decisions, health system operations and more. Furthermore, assessment of immunity in patients with minimal or symptom free infections will provide rich knowledge to assess if certain patients need further risk mitigations (masks, distancing) and which may be safely return to more normal activities.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age; COVID-19 by RT-PCR SARS-CoV-2 assay. (Phase I)

Exclusion Criteria:

* Subjects who tested for COVID-19, but have no available serum specimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 500, but up to 1000 subjects will be enrolled from a retrospective data review and a laboratory information system (LIS) SunQuest identification of COVID-19 (RT-PCR SARS CoV-2) samples.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of antibodies to SARS-CoV-2 | 12 months
  Assessment of prevalence of antibodies to SARS-CoV-2 in subjects tested positive by RT-PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided